CLINICAL TRIAL: NCT05313243
Title: Phase 2 Study of Pembrolizumab and Brentuximab Vedotin in Subjects With Relapsed/Refractory CD30 Positive T-cell Lymphoma
Brief Title: Pembrolizumab and Brentuximab Vedotin in Subjects With Relapsed/Refractory T-cell Lymphoma
Status: Recruiting | Phase: Phase 2 | Type: Interventional
Sponsor: Yale University (Other)
Collaborators: Merck Sharp & Dohme LLC (Industry)
Responsible Party: Principal Investigator, Tarsheen Sethi, MD, MSCI, Assistant Professor of Medicine, Yale University
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: 2000029793; No NIH funding (Other: 11.16.23)
Record Dates: First submitted 2022-03-28; First posted 2022-04-06 (Actual); Last update posted 2025-03-20 (Actual); Status verified 2025-03

CONDITIONS: T-Cell Lymphoma
Keywords: Relapsed; Refractory; CD30 positive; Peripheral T-cell lymphoma; Cutaneous T-cell lymphoma; Pembrolizumab; Brentuximab
MeSH Terms: conditions — Lymphoma, T-Cell; Recurrence; Lymphoma, T-Cell, Peripheral; Lymphoma, T-Cell, Cutaneous | interventions — Brentuximab Vedotin; pembrolizumab

STUDY DESIGN:
Intervention Model Description: All subjects are scheduled to receive up to 16 cycles of combinatorial treatment with brentuximab + pembrolizumab, followed by up to 19 additional cycles of pembrolizumab monotherapy
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: Yes | FDA-regulated Device: No | US Export: No

ARMS (1):
- Brentuximab vedotin (brentuximab) and pembrolizumab (Experimental): All subjects are scheduled to receive up to 16 cycles of combinatorial treatment with brentuximab + pembrolizumab, followed by up to 19 additional cycles of pembrolizumab monotherapy.
  After receiving 35 total doses of pembrolizumab (i.e. scheduled for 16 doses in the combinatorial setting and 8 doses as monotherapy), a subject's pembrolizumab treatment will be complete.
  Interventions: Drug: Brentuximab vedotin; Drug: Pembrolizumab

INTERVENTIONS:
Drug: Brentuximab vedotin — Brentuximab vedotin is an antibody-drug conjugate medication used to treat relapsed or refractory Hodgkin lymphoma (HL) and systemic anaplastic large cell lymphoma (ALCL), a type of T cell non-Hodgkin lymphoma. It selectively targets tumor cells expressing the CD30 antigen, a defining marker of Hodgkin lymphoma and ALCL.
  Other Names: Adcetris
Drug: Pembrolizumab — Pembrolizumab is a humanized antibody used in cancer immunotherapy that treats melanoma, lung cancer, head and neck cancer, Hodgkin lymphoma, stomach cancer, cervical cancer, and certain types of breast cancer.
  Other Names: Keytruda

SUMMARY:
This is a single arm, open label, multicenter study phase 2 study of pembrolizumab and brentuximab in subjects with relapsed/refractory CD30 positive T-cell lymphoma (including peripheral T-cell lymphoma and cutaneous T-cell lymphoma) who have received at least one prior therapy. We hypothesize that this combination is effective and will produce an overall response rate of ~55%. Pembrolizumab and brentuximab will be administered for 16 cycles in subjects with responsive disease. Pembrolizumab will be continued for an additional 19 cycles (total 35 cycles). Response assessments will occur at pre-specified intervals. For the primary endpoint the response assessment after 3 cycles will be taken into consideration. Dose adjustments for specific toxicities with either drug are detailed in the protocol. Based on statistical analysis 32 subjects will need to be accrued to evaluate for disease response based on historical control.

DETAILED DESCRIPTION:
CD30- Positive Peripheral T cell (PTCL) and Cutaneous T cell Lymphomas (CTCL):

T-cell Non-Hodgkin Lymphoma (NHL) includes a clinically heterogeneous group of mature T-cell lymphomas accounting for 10-12% of all NHL. Peripheral T- cell Lymphoma (PTCL) present with clinically aggressive disease with a poor outcome [with the exception of ALK+ Anaplastic Large Cell Lymphomas (ALCL)] and patients experience a high incidence of relapsed/ refractory disease that poses a therapeutic challenge. Despite progress in the past decade in understanding the biology of T-cell lymphomas, with the use of next generation sequencing and molecular profiling of archived tissue samples, there is yet an unmet need in therapeutic options. Amidst the wide range of T-cell lymphoma histologies, PTCL NOS is the most common histological subtype followed by ALCL, angioimmunoblastic lymphoma (AITL) and cutaneous T-cell lymphoma (CTCL). The other histological subtypes (Enteropathy associated T-cell Lymphoma, hepatosplenic T cell lymphoma, NK/T cell lymphoma etc.) account for <5% of T-cell subtypes. Unfortunately, the rare subtypes of T-cell Lymphoma are usually excluded from later phase trials due to their dismal prognosis.

Therapeutic Challenge in Relapsed/ Refractory PTCL and CTCL:

For patients with disease relapse following upfront chemotherapy, stem cell transplantation (SCT) is an option. However, this type of aggressive approach is only feasible in a minority of patients. Despite the advances in the therapeutic arsenal, most of these agents have a modest response rate of 20-30%. More than half of these patients who do respond initially, will ultimately relapse. Conventional chemotherapy in combination with novel agents has been under clinical evaluation with minor improvements in response rates compared with historical controls. Therefore, the urge to optimize therapy by incorporating newer treatments such as novel agents that have a more targeted approach continues to be critically important.

CTCL presents as a chronic disease with a poor prognosis in advanced stage disease. While recently approved agents have expanded the treatment repertoire for CTCL, there is still a need for additional agents as median response with current options averaging about a year(1).

In this context, the efficacy of the novel combination of CD30 directed antibody Brentuximab and PD-1 inhibitor Pembrolizumab in PTCL and CTCL is not known.

ELIGIBILITY:
Inclusion Criteria:

1. Male/female participants who are at least 18 years of age on the day of signing informed consent with histologically confirmed diagnosis of T-cell Non-Hodgkin lymphoma (T-NHL) will be enrolled in this study.
2. The participant (or legally acceptable representative if applicable) provides written informed consent for the trial.
3. Eastern Cooperative Oncology Group (ECOG) performance status of 0-1.
4. Histologically confirmed T-cell Non-Hodgkin lymphoma (T-NHL), including:

   * Peripheral T-cell lymphoma not other specified (PTCL nos)
   * Angioimmunoblastic T-cell lymphoma (AITL)
   * Anaplastic large-cell lymphoma (ALCL)
   * Natural killer (NK)/T-cell lymphoma (nodal or extranodal)
   * Cutaneous T-cell lymphoma (CTCL), including mycosis fungoides (MF)/sezary syndrome
   * Transformed T-cell lymphoma
   * Enteropathy-associated T-cell lymphoma (EATL);
   * Subcutaneous panniculitis-like T-cell lymphoma (SCPTCL)
   * Hepatosplenic T- cell lymphomas.
5. Presence of CD30 (>1%) by IHC on a previous biopsy sample
6. Relapsed/refractory disease having failed at least one prior systemic therapy Note: Single agent Brentuximab could have been a prior line of therapy EXCEPT those with ≥ grade 2 side effects leading to treatment discontinuation or those refractory to Brentuximab
7. For patients with peripheral T-cell lymphoma (PTCL): At least one measurable target lesion ≥1.5 cm
8. A female participant is eligible to participate if she is not pregnant, not breastfeeding, and at least one of the following conditions applies:

   * Not a woman of childbearing potential (WOCBP)
   * A woman of childbearing potential (WOCBP) must have a negative serum or urine pregnancy test during screening within 72 hours prior to receiving first dose of protocol-indicated treatment, and must agree to follow instructions for using acceptable contraception from the time of signing consent, and at least 120 days (4 months) after her final dose of pembrolizumab.
9. A male participant must agree to use contraception during the treatment period and for at least at least 120 days (4 months) after the final dose of pembrolizumab. and refrain from donating sperm during this period.
10. Adequate organ and bone marrow function resulted ≤ 10 days prior to first dose of protocol-indicated treatment:

Exclusion Criteria:

1. Prior therapy with an anti-PD-1, anti-PD-L1, or anti PD L2 agent or with an agent directed to another stimulatory or co-inhibitory T-cell receptor (eg, CTLA-4, OX 40, CD137).
2. Patients with adult T-cell leukemia/ lymphoma (ATLL)
3. Has received prior systemic anti-cancer therapy including investigational agents ≤ 4 weeks prior to first dose of study treatment on Cycle 1, Day 1. Could consider shorter interval for kinase inhibitors or other short half-life drugs.

   Note: concurrent use of bexarotene or vorinostat (where the dose has been stable for the 8 weeks prior to initiating therapy on trial) is permitted for CTCL. Concurrent use of topical steroids or therapies for CTCL is allowed.

   Participants must have recovered from all AEs due to previous therapies to ≤ Grade 1 or to baseline value (i.e. condition prior to initiation of the therapy associated with the AE). Participants with ≤Grade 2 neuropathy as AE may be eligible.

   If participant received major surgery, they must have recovered adequately from the toxicity and/or complications from the intervention prior to starting study treatment.
4. Pregnant or breast-feeding females. A WOCBP who has a positive urine pregnancy test at screening. If the urine test is positive or cannot be confirmed as negative, a serum pregnancy test will be required. In the event that 72 hours have elapsed between the screening pregnancy test and the first dose of study treatment, another pregnancy test (urine or serum) must be performed and must be negative in order for subject to start receiving study medication.
5. Has received radiotherapy within 2 weeks of start of study treatment. Participants must have recovered from all radiation-related toxicities, and not have had radiation pneumonitis. A 1-week washout is permitted for palliative radiation (≤2 weeks of radiotherapy) to non-CNS disease.
6. Has a history of (non-infectious) pneumonitis/interstitial lung disease that required steroids or has current pneumonitis/interstitial lung disease.
7. Has received a live vaccine or live-attenuated vaccine within 30 days prior to the first dose of study drug. Administration of killed vaccines is allowed.
8. Is currently participating in or has participated in a study of an investigational agent or has used an investigational device within 4 weeks prior to the first dose of study treatment.

   Note: Participants who have entered the follow-up phase of an investigational study may participate as long as it has been 4 weeks after the last dose of the previous investigational agent.
9. Has a diagnosis of immunodeficiency or is receiving chronic systemic steroid therapy (in dosing exceeding 10 mg daily of prednisone equivalent) or any other form of immunosuppressive therapy within 7 days prior to the first dose of study drug.
10. Has active autoimmune disease that has required systemic treatment in the past one year (i.e. with use of disease modifying agents, corticosteroids or immunosuppressive drugs).

    Replacement therapy (eg., thyroxine, insulin, or physiologic corticosteroid replacement therapy for adrenal or pituitary insufficiency, etc.) is not considered a form of systemic treatment. Subjects with type I diabetes mellitus, hypothyroidism only requiring hormone replacement, skin disorders (such as vitiligo, psoriasis or alopecia) not requiring systemic treatment, or conditions not expected to recur in the absence of an external trigger are permitted to enroll.
11. Active uncontrolled infection requiring systemic therapy (patients must be afebrile for ≥ 48 hours off antibiotics prior to first protocol treatment). If fever is attributed to tumor fever (B symptom) then this criteria would not apply.
12. Active myocarditis, regardless of etiology; or New York Heart Association (NYHA) functional classification III-IV heart failure.
13. Known active CNS metastases and/or carcinomatous meningitis. Participants with previously treated brain metastases may participate provided they are radiologically stable, i.e. without evidence of progression for at least 4 weeks by repeat imaging (note that the repeat imaging should be performed during study screening), clinically stable and without requirement of steroid treatment for at least 14 days prior to first dose of study treatment.
14. Disease free of prior malignancies for ≥ 1 year with exception of currently treated basal cell or squamous cell carcinoma of the skin, or carcinoma "in situ" of the cervix or breast. (Other malignancies will require advance discussion and agreement between the investigator and the sponsor-investigator regarding risk of recurrence.)
15. Known severe hypersensitivity (≥Grade 3) to pembrolizumab and/or any of its excipients.
16. Has a known history of Human Immunodeficiency Virus (HIV). Note: No HIV testing is required unless mandated by local health authority.
17. Has a known history of Hepatitis B (defined as Hepatitis B surface antigen [HBsAg] reactive) or known active Hepatitis C virus (defined as HCV RNA [qualitative] is detected) infection. Note: no testing for Hepatitis B and Hepatitis C is required unless mandated by local health authority.
18. Has a history or current evidence of any condition (e.g. renal disease that would preclude treatment or obstructive pulmonary disease and history of bronchospasm), therapy, or laboratory abnormality that might confound the results of the study, interfere with the subject's participation for the full duration of the study, or is not in the best interest of the subject to participate, in the opinion of the treating investigator.
19. Clinically significant history of liver disease, including current alcohol abuse or cirrhosis.
20. Known psychiatric or substance abuse disorders that would interfere with cooperation with the requirements of the trial.
21. Has a known history of active TB (Bacillus Tuberculosis).
22. Prior allogeneic stem cell transplant within last 5 years or active graft vs. host disease (GVHD).
23. Patients with grade 2 or higher peripheral neuropathy

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 32 (Estimated)
Dates: Start 2023-07-10 (Actual); Primary Completion 2028-04-30 (Estimated); Study Completion 2028-07-30 (Estimated)

PRIMARY OUTCOMES:
The best overall response with the combination of brentuximab and pembrolizumab. | 3 cycles (63 Days)
  As assessed by the Lugano criteria for PTCL(16) and the global response score for CTCL(17)

SECONDARY OUTCOMES:
Occurrence of toxicity | 2 Years
  As assessed by using the NCI Common Terminology Criteria for Adverse Events version 5 (CTCAE v5) for grading
Progression free survival (PFS) | 2 Years
  Defined as the time from enrollment to earliest of progression, death or follow-up
Overall survival (OS) | 2 Years
  Defined as the time from enrollment to death or last follow-up
Time to treatment failure | 2 Years
  Defined as interval from initiation of chemotherapy to premature discontinuation for any reason.
Duration of response | 2 Years
  Defined as the interval from response initiation (when either CR or PR is first determined) to progression or death, whichever occurs first.
Time to progression | 2 Years
  Defined as the time from treatment initiation to tumor progression.

CONTACTS AND LOCATIONS:
Overall Officials: Tarsheen Sethi, MD, Principal Investigator — Yale University
Locations (2):
- United States (2):
  - Yale Smilow Cancer Hospital, New Haven, Connecticut
  - Dana Farber Cancer Institute, Boston, Massachusetts

REFERENCES:
- [Background] Prince HM, Kim YH, Horwitz SM, Dummer R, Scarisbrick J, Quaglino P, Zinzani PL, Wolter P, Sanches JA, Ortiz-Romero PL, Akilov OE, Geskin L, Trotman J, Taylor K, Dalle S, Weichenthal M, Walewski J, Fisher D, Dreno B, Stadler R, Feldman T, Kuzel TM, Wang Y, Palanca-Wessels MC, Zagadailov E, Trepicchio WL, Zhang W, Lin HM, Liu Y, Huebner D, Little M, Whittaker S, Duvic M; ALCANZA study group. Brentuximab vedotin or physician's choice in CD30-positive cutaneous T-cell lymphoma (ALCANZA): an international, open-label, randomised, phase 3, multicentre trial. Lancet. 2017 Aug 5;390(10094):555-566. doi: 10.1016/S0140-6736(17)31266-7. Epub 2017 Jun 7. PMID 28600132
- [Background] Mohammed HO, Yamamoto R, Carpenter TE, Ortmayer HB. Comparison of egg yolk and serum for the detection of Mycoplasma gallisepticum and M. synoviae antibodies by enzyme-linked immunosorbent assay. Avian Dis. 1986 Apr-Jun;30(2):398-408. PMID 3729886
- [Background] Gunraj DR, Rajapakse DA. Daily ECG confirmation in acute myocardial infarction. Practitioner. 1974 Sep;213(1275):361-4. No abstract available. PMID 4425442
- [Background] Wartewig T, Kurgyis Z, Keppler S, Pechloff K, Hameister E, Ollinger R, Maresch R, Buch T, Steiger K, Winter C, Rad R, Ruland J. PD-1 is a haploinsufficient suppressor of T cell lymphomagenesis. Nature. 2017 Dec 7;552(7683):121-125. doi: 10.1038/nature24649. Epub 2017 Nov 15. PMID 29143824
- [Background] Connor AM, Moshiri F. Advancement genioplasty: an important part of combination surgery in black American patients. Am J Orthod Dentofacial Orthop. 1988 Feb;93(2):92-8. doi: 10.1016/0889-5406(88)90285-5. No abstract available. PMID 3422534
- [Background] Gerdes MJ, Sevinsky CJ, Sood A, Adak S, Bello MO, Bordwell A, Can A, Corwin A, Dinn S, Filkins RJ, Hollman D, Kamath V, Kaanumalle S, Kenny K, Larsen M, Lazare M, Li Q, Lowes C, McCulloch CC, McDonough E, Montalto MC, Pang Z, Rittscher J, Santamaria-Pang A, Sarachan BD, Seel ML, Seppo A, Shaikh K, Sui Y, Zhang J, Ginty F. Highly multiplexed single-cell analysis of formalin-fixed, paraffin-embedded cancer tissue. Proc Natl Acad Sci U S A. 2013 Jul 16;110(29):11982-7. doi: 10.1073/pnas.1300136110. Epub 2013 Jul 1. PMID 23818604
- [Background] McKinley ET, Sui Y, Al-Kofahi Y, Millis BA, Tyska MJ, Roland JT, Santamaria-Pang A, Ohland CL, Jobin C, Franklin JL, Lau KS, Gerdes MJ, Coffey RJ. Optimized multiplex immunofluorescence single-cell analysis reveals tuft cell heterogeneity. JCI Insight. 2017 Jun 2;2(11):e93487. doi: 10.1172/jci.insight.93487. eCollection 2017 Jun 2. PMID 28570279
- [Background] Byford ET, Carr M, Ladikou E, Ahearne MJ, Wagner SD. Circulating Tfh1 (cTfh1) cell numbers and PD1 expression are elevated in low-grade B-cell non-Hodgkin's lymphoma and cTfh gene expression is perturbed in marginal zone lymphoma. PLoS One. 2018 Jan 2;13(1):e0190468. doi: 10.1371/journal.pone.0190468. eCollection 2018. PMID 29293620
- [Background] Leelatian N, Diggins KE, Irish JM. Characterizing Phenotypes and Signaling Networks of Single Human Cells by Mass Cytometry. Methods Mol Biol. 2015;1346:99-113. doi: 10.1007/978-1-4939-2987-0_8. PMID 26542718
- [Background] Oken MM, Creech RH, Tormey DC, Horton J, Davis TE, McFadden ET, Carbone PP. Toxicity and response criteria of the Eastern Cooperative Oncology Group. Am J Clin Oncol. 1982 Dec;5(6):649-55. No abstract available. PMID 7165009
- [Background] Cockcroft DW, Gault MH. Prediction of creatinine clearance from serum creatinine. Nephron. 1976;16(1):31-41. doi: 10.1159/000180580. PMID 1244564
- [Background] Weisenburger DD, Savage KJ, Harris NL, Gascoyne RD, Jaffe ES, MacLennan KA, Rudiger T, Pileri S, Nakamura S, Nathwani B, Campo E, Berger F, Coiffier B, Kim WS, Holte H, Federico M, Au WY, Tobinai K, Armitage JO, Vose JM; International Peripheral T-cell Lymphoma Project. Peripheral T-cell lymphoma, not otherwise specified: a report of 340 cases from the International Peripheral T-cell Lymphoma Project. Blood. 2011 Mar 24;117(12):3402-8. doi: 10.1182/blood-2010-09-310342. Epub 2011 Jan 26. PMID 21270441
- [Background] Pro B, Advani R, Brice P, Bartlett NL, Rosenblatt JD, Illidge T, Matous J, Ramchandren R, Fanale M, Connors JM, Fenton K, Huebner D, Pinelli JM, Kennedy DA, Shustov A. Five-year results of brentuximab vedotin in patients with relapsed or refractory systemic anaplastic large cell lymphoma. Blood. 2017 Dec 21;130(25):2709-2717. doi: 10.1182/blood-2017-05-780049. Epub 2017 Oct 3. PMID 28974506
- [Background] Wilcox RA, Feldman AL, Wada DA, Yang ZZ, Comfere NI, Dong H, Kwon ED, Novak AJ, Markovic SN, Pittelkow MR, Witzig TE, Ansell SM. B7-H1 (PD-L1, CD274) suppresses host immunity in T-cell lymphoproliferative disorders. Blood. 2009 Sep 3;114(10):2149-58. doi: 10.1182/blood-2009-04-216671. Epub 2009 Jul 13. PMID 19597183
- [Background] Chen BJ, Chapuy B, Ouyang J, Sun HH, Roemer MG, Xu ML, Yu H, Fletcher CD, Freeman GJ, Shipp MA, Rodig SJ. PD-L1 expression is characteristic of a subset of aggressive B-cell lymphomas and virus-associated malignancies. Clin Cancer Res. 2013 Jul 1;19(13):3462-73. doi: 10.1158/1078-0432.CCR-13-0855. Epub 2013 May 14. PMID 23674495
- [Background] Kwong YL, Chan TSY, Tan D, Kim SJ, Poon LM, Mow B, Khong PL, Loong F, Au-Yeung R, Iqbal J, Phipps C, Tse E. PD1 blockade with pembrolizumab is highly effective in relapsed or refractory NK/T-cell lymphoma failing l-asparaginase. Blood. 2017 Apr 27;129(17):2437-2442. doi: 10.1182/blood-2016-12-756841. Epub 2017 Feb 10. PMID 28188133
- [Background] Barta SK, Zain J, MacFarlane AW 4th, Smith SM, Ruan J, Fung HC, Tan CR, Yang Y, Alpaugh RK, Dulaimi E, Ross EA, Campbell KS, Khan N, Siddharta R, Fowler NH, Fisher RI, Oki Y. Phase II Study of the PD-1 Inhibitor Pembrolizumab for the Treatment of Relapsed or Refractory Mature T-cell Lymphoma. Clin Lymphoma Myeloma Leuk. 2019 Jun;19(6):356-364.e3. doi: 10.1016/j.clml.2019.03.022. Epub 2019 Apr 3. PMID 31029646
- [Background] Cheson BD, Ansell S, Schwartz L, Gordon LI, Advani R, Jacene HA, Hoos A, Barrington SF, Armand P. Refinement of the Lugano Classification lymphoma response criteria in the era of immunomodulatory therapy. Blood. 2016 Nov 24;128(21):2489-2496. doi: 10.1182/blood-2016-05-718528. Epub 2016 Aug 29. PMID 27574190
- [Background] Cheson BD, Fisher RI, Barrington SF, Cavalli F, Schwartz LH, Zucca E, Lister TA; Alliance, Australasian Leukaemia and Lymphoma Group; Eastern Cooperative Oncology Group; European Mantle Cell Lymphoma Consortium; Italian Lymphoma Foundation; European Organisation for Research; Treatment of Cancer/Dutch Hemato-Oncology Group; Grupo Espanol de Medula Osea; German High-Grade Lymphoma Study Group; German Hodgkin's Study Group; Japanese Lymphorra Study Group; Lymphoma Study Association; NCIC Clinical Trials Group; Nordic Lymphoma Study Group; Southwest Oncology Group; United Kingdom National Cancer Research Institute. Recommendations for initial evaluation, staging, and response assessment of Hodgkin and non-Hodgkin lymphoma: the Lugano classification. J Clin Oncol. 2014 Sep 20;32(27):3059-68. doi: 10.1200/JCO.2013.54.8800. PMID 25113753
- [Background] Herbaux C, Merryman R, Devine S, Armand P, Houot R, Morschhauser F, Haverkos B. Recommendations for managing PD-1 blockade in the context of allogeneic HCT in Hodgkin lymphoma: taming a necessary evil. Blood. 2018 Jul 5;132(1):9-16. doi: 10.1182/blood-2018-02-811174. Epub 2018 May 2. PMID 29720488